CLINICAL TRIAL: NCT00749775
Title: Eplerenone Observational Study Of Safety And Efficacy Evaluation To Normalize Blood Pressure For Clinical Effectiveness
Brief Title: Selara Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Acronym: ESSENCE
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6141113
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
Keywords: Eplerenone; Selara; Hypertension; Good post-marketing study Practice; Drug use Investigation; Regulatory Post Marketing Commitment Plan; ESSENCE
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eplerenone: Subjects who are treated with Eplerenone tablet for hypertension disease
  Interventions: Drug: Selara

INTERVENTIONS:
Drug: Selara — Treatment should be initiated at 25 mg once daily and titrated to the recommended dose of 50 mg once daily, preferably within 4 weeks as tolerated by the patient. Selara may be administered with or without food.

SUMMARY:
To collect the efficacy and safety information of Eplerenone on patients with hypertension related to their appropriate use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients who are prescribed Selara tablet for Hypertension.

Exclusion Criteria:

* Subjects who have been prescribed Selara tablet.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6141113 prescribes the Selara tablet.
Sampling Method: Probability Sample
Enrollment: 3338 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141113&StudyName=Selara%20Drug%20use%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Selara: Participants taking Selara according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Selara
Started | 3317
Completed | 3210
Not Completed | 107
Not completed — Protocol Violation | 24
Not completed — Lost to Follow-up | 36
Not completed — No visit after first day of treatment | 44
Not completed — No drug administration | 3

BASELINE CHARACTERISTICS:
Arm/Group | Selara
Number analyzed (Participants) | 3210
Age, Customized [Number; unit: participants]
  <65 years old | 1224
  >=65 years old | 1986
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1539
  Male | 1671

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Selara, irrespective of causal relationship to Selara (including clinically problematic abnormal changes in laboratory test values). Treatment Related Adverse Events were evaluated in company with the causal relationship to Selara.
Time Frame: 12 weeks
Population: No statistical analysis provided for the frequency of Treatment Related adverse events.
Measure: Number; unit: participants
Arm/Group | Selara
Number analyzed (Participants) | 3210
participants | 75

2. Primary Outcome: Number of Participants With Serious Treatment Related Adverse Events.
Description: Serious treatment related adverse events mean those that may lead to death, life-threatening, hospitalization or prolonged hospitalization, a permanent or remarkable disorder/dysfunction, congenital anomaly/congenital deficiency, or other medically significant events or disorder.
Time Frame: 12 weeks
Population: No statistical analysis provided for the frequency of serious treatment related adverse events.
Measure: Number; unit: participants
Arm/Group | Selara
Number analyzed (Participants) | 3210
participants | 16

3. Secondary Outcome: Change in Systolic Blood Pressure Over Time.
Description: The primary analysis item was the mean systolic blood pressure at 4, 8, and 12 weeks of the observation period or at last evaluation date if Selara was terminated prematurely.
Time Frame: 12 weeks
Population: The efficacy analysis population basically consists of the evaluable participants in accordance with the separately prepared analysis plan (participants judged to have been evaluated appropriately).
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- At Baseline: Mean systolic blood pressure at baseline among Participants taking Selara according to Japanese Package Insert.
- At 4 Weeks: Mean systolic blood pressure at 4 weeks among Participants taking Selara according to Japanese Package Insert.
- At 8 Weeks: Mean systolic blood pressure at 8 weeks among Participants taking Selara according to Japanese Package Insert.
- At 12 Weeks: Mean systolic blood pressure at 12 weeks among Participants taking Selara according to Japanese Package Insert.
- At Last Evaluation Date: Mean systolic blood pressure at last evaluation date among Participants taking Selara according to Japanese Package Insert.
Arm/Group | At Baseline | At 4 Weeks | At 8 Weeks | At 12 Weeks | At Last Evaluation Date
Number analyzed (Participants) | 2252 | 880 | 756 | 730 | 2150
mmHg | 151.8 (19.6) | 140.7 (17.7) | 137.5 (16.2) | 134.7 (15.6) | 134.0 (15.9)
Statistical Analysis 1: Comparison: At Baseline vs At 4 Weeks; The null hypothesis is that the mean systolic blood pressure at 4 weeks does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: At Baseline vs At 8 Weeks; The null hypothesis is that the mean systolic blood pressure at 8 weeks does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 3: Comparison: At Baseline vs At 12 Weeks; The null hypothesis is that the mean systolic blood pressure at 12 weeks does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 4: Comparison: At Baseline vs At Last Evaluation Date; The null hypothesis is that the mean systolic blood pressure at last evaluation date does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis

4. Secondary Outcome: Change in Diastolic Blood Pressure Over Time.
Description: The primary analysis item was the mean diastolic blood pressure at 4, 8, and 12 weeks of the observation period or at last evaluation date if Selara was terminated prematurely.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- At Baseline: Mean diastolic blood pressure at baseline among Participants taking Selara according to Japanese Package Insert.
- At 4 Weeks: Mean diastolic blood pressure at 4 weeks among Participants taking Selara according to Japanese Package Insert.
- At 8 Weeks: Mean diastolic blood pressure at 8 weeks among Participants taking Selara according to Japanese Package Insert.
- At 12 Weeks: Mean diastolic blood pressure at 12 weeks among Participants taking Selara according to Japanese Package Insert.
- At Last Evaluation Date: Mean diastolic blood pressure at last evaluation date among Participants taking Selara according to Japanese Package Insert.
Arm/Group | At Baseline | At 4 Weeks | At 8 Weeks | At 12 Weeks | At Last Evaluation Date
Number analyzed (Participants) | 2252 | 880 | 756 | 730 | 2150
mmHg | 85.1 (13.9) | 79.5 (12.9) | 78.0 (12.5) | 76.6 (11.8) | 77.0 (11.7)
Statistical Analysis 1: Comparison: At Baseline vs At 4 Weeks; The null hypothesis is that the mean diastolic blood pressure at 4 weeks does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: At Baseline vs At 8 Weeks; The null hypothesis is that the mean diastolic blood pressure at 8 weeks does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 3: Comparison: At Baseline vs At 12 Weeks; The null hypothesis is that the mean diastolic blood pressure at 12 weeks does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 4: Comparison: At Baseline vs At Last Evaluation Date; The null hypothesis is that the mean diastolic blood pressure at last evaluation date does not differ from that at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis

5. Secondary Outcome: Number of Participants That Responded to Selara Treatment.
Description: Number of participants among the efficacy analysis population that responded to Selara treatment.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Selara
Number analyzed (Participants) | 3009
participants | 2772

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The frequency of treatment related adverse events during the study.
Arm/Group | Selara
Serious Adverse Events (participants affected / at risk) | 16/3210
Other Adverse Events (participants affected / at risk) | 59/3210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selara (N=3210)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3)
Drug interaction (General disorders) | 1 (1)
Blood potassium increased (Investigations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selara (N=3210)
Herpes zoster (Infections and infestations) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Convulsion (Nervous system disorders) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 4 (4)
Polyuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 4 (4)
Blood creatinine increased (Investigations) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.